CLINICAL TRIAL: NCT06354166
Title: Contribution of a Digital Tool Combined With Supportive Human Coordination for Transitional Care of Patients in Unscheduled Hospitalisation in Geriatric Short-stay Care
Brief Title: Study Human Digital Support Transitional Care
Acronym: SUNH-ST
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Divoluci (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2023-A02745-40
Record Dates: First submitted 2024-04-03; First posted 2024-04-09 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Aging

STUDY DESIGN:
Intervention Model Description: Interventional, randomised (1:1 ratio), single-centre study
Masking Description: open-label study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Divomed digital tool combined with human coordination (Experimental): A digital tool combined with human coordination (Divomed) to organise discharge home from the start of hospitalisation. The digital application will be interconnected with the patient's medical file.
  Interventions: Procedure: Unscheduled hospital admissions
- Control Group (Active Comparator): The control group corresponds to the organisation of conventional hospital discharge from the geriatric short-stay department.
  The digital application will be interconnected with the patient's medical file.
  Interventions: Procedure: Unscheduled hospital admissions

INTERVENTIONS:
Procedure: Unscheduled hospital admissions — Unscheduled short-stay geriatric hospitalisations of people aged over 75 to their homes

SUMMARY:
The purpose of the study is to compare the effectiveness of Divomed in organising complex hospital discharges with a conventional organisation. Effectiveness will be assessed by reducing the length of stay of patients in geriatric short-stay care.

DETAILED DESCRIPTION:
This is an interventional, randomised (ratio 1:1), single-centre, open-label study evaluating Divomed, a digital tool combined with human coordination, to speed up the discharge of people aged over 75 from unscheduled short-stay geriatric hospital admissions to their homes.

The study population will be patients aged 75 or over, admitted for short term unscheduled geriatric hospitalisation and eligible for discharge home.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 75 years ;
* Unplanned hospitalisation from emergency, transfers from other inpatient departments or outpatient medicine;
* Patient eligible for short-stay geriatric hospitalisation estimated to last at least 10 days;
* Patient eligible for a return home;
* Patients who have been informed and have signed an informed consent form. If necessary (for cognitive or other reasons), the information must be given to a third party, i.e. the patient's legal representative or trusted person (independent of the investigator and the sponsor), who may be asked to sign or co-sign the informed consent form (depending on the patient's vulnerability).

Exclusion Criteria:

* Patients scheduled for transfusion, iron infusion or colonoscopy;
* Patients in palliative care;
* Geographical area other than department 37;
* Planned discharge from hospital to a residential establishment for dependent elderly people or to follow-up and rehabilitation care or long-term care units;
* Patient or deprived of liberty by judicial or administrative decision ;
* Patient participating in or being excluded from another clinical trial;
* Patients not covered by a social security scheme.

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
length of stay | 1 month
  The effectiveness of Divomed in organising complex hospital discharges will be assessed at discharge by comparing lengths of stay in the 2 groups.

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU de Tours - Hôpital Bretonneau, Tours, France